CLINICAL TRIAL: NCT00105755
Title: Dermal Thermometry and Self-Care of High Risk Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IIR 20-059
Record Dates: First submitted 2005-03-16; First posted 2005-03-17 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Diabetes Mellitus; Ulcer; Diabetic Polyneuropathy
Keywords: Activity Cycles; Amputation; Prevention; Temperature
MeSH Terms: conditions — Diabetes Mellitus; Ulcer; Diabetic Neuropathies | interventions — Equipment and Supplies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Device: personal dermal thermometer (DT); Device: Device

INTERVENTIONS:
Device: personal dermal thermometer (DT)
Device: Device

SUMMARY:
Foot ulcers remain the most common reason for hospital admission among veterans with diabetes. Healing and preventing these wounds should be a high priority for clinicians treating these high-risk patients. Previous work by the investigators has suggested that diabetic foot ulcers are preceded by inflammation, which can potentially be detected with a thermometer.

DETAILED DESCRIPTION:
Background:

Foot ulcers remain the most common reason for hospital admission among veterans with diabetes. Healing and preventing these wounds should be a high priority for clinicians treating these high-risk patients. Previous work by the investigators has suggested that diabetic foot ulcers are preceded by inflammation, which can potentially be detected with a thermometer.

Objectives:

The purpose of this project is to evaluate the utility of a novel personal dermal thermometry system to empower patients and caregivers and thereby reduce the risk for lower extremity ulceration and amputation in veterans at high risk for these complications.

Methods:

In this randomized clinical trial, 384 patients are being enrolled and assigned to either standard of care (SC) or SC plus a personal dermal thermometer (DT) to evaluate and log their plantar skin temperatures. All patients are given access to a 24 hour "hot foot line" to call for immediate access to care if they identify a hot spot (DT group) or a site of concern on standard self-evaluation (SC). All patients are assigned a sophisticated computerized activity monitor, which allows investigators access to time and magnitude of activity, downloaded at regular patient visits.

Status:

Project work is complete

ELIGIBILITY:
Inclusion Criteria:

vibration perception threshold needs to be greater than 25, palpable pulse, Over 18 years of age Has Diabetes and Neuropathy

Exclusion Criteria:

No ulcers. Unable to walk without assistance of wheelchair or crutches

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2003-01; Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Reduce the risk for lower extremity ulceration and amputation in veterans at high risk for these complications.; Incidence of diabetic foot ulcers over 18 months. Incidence of foot infections over 18 months. Incidence of Charcot fractures.

SECONDARY OUTCOMES:
Improve quality of life. Health Related Quality of Life (change over 18 months)

CONTACTS AND LOCATIONS:
Overall Officials: Brent Nixon, DPM MBA BA, Principal Investigator — Southern Arizona VA Health Care System, Tucson, AZ
Locations (1):
- Southern Arizona VA Health Care System, Tucson, AZ, Tucson, Georgia, United States

REFERENCES:
- [Result] Armstrong DG, Lavery LA, Holtz-Neiderer K, Mohler MJ, Wendel CS, Nixon BP, Boulton AJ. Variability in activity may precede diabetic foot ulceration. Diabetes Care. 2004 Aug;27(8):1980-4. doi: 10.2337/diacare.27.8.1980. PMID 15277427
- [Derived] Armstrong DG, Holtz-Neiderer K, Wendel C, Mohler MJ, Kimbriel HR, Lavery LA. Skin temperature monitoring reduces the risk for diabetic foot ulceration in high-risk patients. Am J Med. 2007 Dec;120(12):1042-6. doi: 10.1016/j.amjmed.2007.06.028. PMID 18060924